CLINICAL TRIAL: NCT06399978
Title: The Feasibility and Effect of Cognitive Training on Objective and Subjective Cognitive Functioning in Patients With Mild Cognitive Impairment: A Pilot Study
Brief Title: The Feasibility and Effect of Digital Cognitive Training in Mild Cognitive Impairment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pernille Louise Kjeldsen (Other)
Collaborators: Brain+ ApS (Unknown); Eurostars EUREKA (Unknown); Innovation Fund Denmark (Individual); University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Pernille Louise Kjeldsen, Project coordinator, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACTTDCS
Record Dates: First submitted 2024-03-20; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Alzheimer's disease; Cognitive functioning; Quality of life; Digital cognitive training; Gamified cognitive training
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: In this study, 40 MCI participants will be randomly assigned to either an intervention group (digital cognitive training with a gamified DOT programme, N=20) or an active control group (digital cognitive training with a gamified non-DOT programme, N=20).
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gamified DOT (Experimental): Participants perform digital cognitive training with a program based on the Differential Outcomes Training (DOT) principle, in which each stimulus-response association to be learnt is followed by a unique reinforcer/outcome, in order to boost associative learning.
  Interventions: Behavioral: Brain Blossom - Gamified Differential Outcome Training
- Gamified non-DOT (Active Comparator): Participants perform digital cognitive training with a non-Differential Outcomes Training (NDOT) programme, in which each stimulus-response association to be learnt is followed by a random reinforcer/outcome.
  Interventions: Behavioral: Gamified Non-Differential Outcome Training

INTERVENTIONS:
Behavioral: Brain Blossom - Gamified Differential Outcome Training — Digital cognitive training with a gamified DOT task for 20 minutes per day 3-4 times a week for 6-8 weeks.
  Other Names: DOT
  Arms: Gamified DOT
Behavioral: Gamified Non-Differential Outcome Training — Digital cognitive training with a gamified NDOT task for 20 minutes per day 3-4 times a week for 6-8 weeks.
  Other Names: NDOT
  Arms: Gamified non-DOT

SUMMARY:
The goal of this study is to assess the feasibility and effect of digital cognitive training based on the principles of Differential Outcome Training (DOT) in patients with Mild Cognitive Impairment. In DOT training, each stimulus-response pair to be learnt is followed by a unique reinforcer, as opposed to non-DOT (NDOT) training, where the stimulus-response pairs are all followed by a random reinforcer. DOT training is believed to boost learning more than NDOT training through associations.

The main questions the study aims to answer are:

* Whether at-home, tablet-based digital cognitive training is feasible in elderly patients with Mild Cognitive Impairment
* Whether regularly digital cognitive DOT training has a positive effect on patients' cognitive functioning and quality of life
* Whether any potential effects that the cognitive DOT training may have on the patients' cognitive functioning are transferable to the patients' daily life.

Participation in the study includes:

* A pre-training session at the site with the primary project coordinator, where the patient will complete a number of self-report questionnaires about their health, cognition, and quality of life as well as a neuropsychological assessment.
* Training with the digital cognitive DOT training program at home for 20 min. per day 3-4 times a week for 6-8 weeks.
* A post-training session at the site with the primary project coordinator after the 6-8 weeks have passed, where the patient will complete a usability questionnaire about the training programme, some of the same self-report questionnaires about their health, cognition, and quality of life as well as some of the neuropsychological assessments.
* A 1-month follow-up session where the patients will complete some of the same self-report questionnaires again about their cognition and quality of life plus a questionnaire aimed the transferability of any positive cognitive effects of the training.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is the most common form of dementia, a debilitating neurodegenerative disease with cognitive impairments, especially impairments in memory, at its core. AD is progressive, with cognitive symptoms gradually worsening as AD brain pathology builds over time. The clinical construct of Mild Cognitive Impairment (MCI) represents an intermediate stage between healthy ageing and early dementia with cognitive impairment that is worse than what is seen in healthy ageing, but not enough to interfere with daily living. Although, not all MCI cases lead to dementia, the majority of cases eventually progress.

The amnestic subtype of MCI, which is especially characterised by the presence of memory impairments, is the most likely to progress to AD dementia. In line with the evolution of brain neurodegeneration in AD, typically beginning in memory-related medial-temporal limbic areas, which specifically contribute to forming and accessing spatial contextual short-term memories, spatial memory deficits are especially common in amnestic MCI. AD patients and even amnestic MCI patients perform worse on visuospatial short-term memory tasks compared to healthy participants and individuals with other neurodegenerative disorders. Memory functions are essential for daily living, and memory impairments have been shown to be a major determinant of health outcomes and well-being in age-related disorders.

At the time an MCI diagnosis is made, the pathological burden is often so high that it is almost impossible to stop or reverse the cognitive impairment. Presently, there is no cure for AD or any other type of dementia, and available pharmacological treatments have only very limited effects on cognitive symptoms. A major research priority should therefore be to develop non-pharmacological approaches, which are cost-effective and potentially feasible for large-scale implementation, to preserve and promote cognitive function and improve quality of life early on in MCI.

Previous studies have shown beneficial effects of cognitive training in MCI and AD patients using a novel training procedure that has been proposed to active and relay on memory processes and brain structures that are less affected in MCI and AD - The Differential Outcome Training (DOT). DOT training is based on the principle that each stimulus-response association to be learned is followed by a unique reinforcer, relative to a condition where reinforcers are presented randomly (non-differential outcomes training, NDOT). DOT training has been shown to result in enhanced learning, including faster acquisition, better overall retention, and higher retention accuracy, in both animals and humans. Nonetheless, the effects of a prolonged DOT training on visuospatial short-term memory performance and possible transfer of any benefits to other memory tasks and cognitive domains as well as its impact on quality of life in patients with MCI requires further research.

This study aims to establish the feasibility and effectiveness of a recently developed digital, gamified type of cognitive training in individuals with MCI. The study aims to address this by using a recently developed gamified version of the DOT task. This gamified DOT task integrates the DOT procedure within a gardening task. Participants are introduced to a botanic garden that they have to keep up, which includes cleaning up, obtaining seeds, planting plants, and putting up decorations. They can obtain seeds, plants, and money by performing a visuospatial short-term memory DOT task, which they can then use for the garden.

The purpose of this study is threefold: 1) to assess if digital, gamified cognitive training at home is feasible in elderly patients with MCI, 2) to explore the effectiveness of the gamified version of the DOT task on MCI patients' cognitive functioning and quality of life, and 3) to explore any possible transfer benefits of the DOT training to other cognitive tasks and to individuals' self-report measures of quality of life.

For this study, 40 MCI patients aged 65-80 will be recruited from the local Dementia Clinic. The patients will be randomly assigned to an intervention group (gamified DOT group, N=20) and an active control group (gamified NDOT, N=20). The patients will meet with the project coordinator for a pre-training session to assess their cognitive functioning and wellbeing prior to the cognitive training, after which they will complete 6-8 weeks of training at home, and will upon completion of the training come back in for a post-training session to assess whether the patients found the cognitive training feasible and whether the training has had an effect on the patients' cognitive functioning and wellbeing.

The study follows the Helsinki Declaration and will not begin before the necessary ethical and other approvals have been obtained. Laws and guidelines regarding handling personal data (GDPR rules) will also be followed with regards to all parts of the study.

ELIGIBILITY:
Inclusion Criteria (MCI patients):

* Age: 65-80
* MCI diagnosis made by a specialist in a Dementia Clinic:

  * Meeting the diagnostic criteria for a diagnosis of MCI
  * Abnormal memory function compared to age and education as assessed with a neuropsychological assessment prior to enrolment in the study
  * Generally preserved Activities of Daily Living (ADL)
  * Not demented
* MCI diagnosis should be made no more than 6 months before enrolment in the study

Exclusion Criteria:

* Significant systemic disease or unstable medical or psychiatric disorder
* Past history of stroke, brain damage, head trauma, or concussion, which significantly affects level of functioning
* Past history of significant alcohol or drug abuse
* Significantly impaired vision or hearing
* Colour blindness
* Danish as a second language
* Participation in any other clinical studies during project participation

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Usability of the digital cognitive training program assessed with a self-report questionnaire | Post-training (6-8 weeks)
  Participants are asked to fill out a self-report questionnaire made specifically for this study. The questionnaire includes 10 questions about the participants' experience with the digital cognitive training post-training, including whether the programme ran smoothly, was easy to use, was engaging, and was fun, and whether the participants would be interested in playing it or similar game again in the future.
Memory task performance assessed with a Differential Outcome Task (DOT task) | Post-training (6-8 weeks)
  Participants are asked to complete a computerised face recognition DOT task. Participants are presented with different faces and asked which ones they have seen previously. The responses are each followed by an outcome. There are two versions of the task: a DOT version where each correctly identified face is associated with a certain outcome, and a NDOT version, in which the outcomes appear randomly.
Visuo-spatial memory task performance assessed with a gamified visuo-spatial memory task (Starry Night) | Post-training (6-8 weeks)
  Participants are asked to complete the 20-min gamified visuo-spatial memory task, Starry Night. Participants are presented with complex patterns somewhere on a screen for a few seconds at a time. After a short pause, different complex patterns appear on the screen, of which one was the pattern the participant just saw. The participant needs to both choose the correct pattern and then place it on the spot on the screen where it previously appeared.
Subjective cognitive functioning assessed by the 20-Item Short-Form Change in Cognition Scale (CCI-S-20) | Post-training (6-8 weeks)
  Participants are asked to fill out the 20-Item Short-Form Change in Cognition Scale (CCI-S-20). This version of the questionnaire contains 20 questions about memory functions in daily life. Participants indicate on a 5-point rating scale if they think their own memory functions are the same as they have always been or if they have become worse, and if so, to which degree. Participants' ratings can be between 0 ('no change in that memory function') to 4 ('severe change in that memory function'). A higher score indicates worse cognition.
Quality of life assessed with the Quality of Life Ladder (QoL Ladder) | Post-training (6-8 weeks)
  The Quality of Life Ladder is a commonly used, simple task. Participants are asked to rate their quality of life on a scale from 1 to 8, where 1 is the worst and 8 is the best possible quality of life they could realistically have.
Depressive symptoms assessed with the 15-Item Geriatric Depression Scale (GDS-15) | Post-training (6-8 weeks)
  Participants are asked to fill out the 15-Item Geriatric Depression scale (GDS-15). The GDS is a very commonly used measure for depressive symptoms in elderly individuals. The participants are presented with 15 yes- or no-questions. Their responses for each question are coded as either 0 or 1, where 0 indicates that depressive symptoms are not present, while a score of 1 indicates the presence of a depressive symptom. Participants can score between 0 and 15, where a higher score indicates worse mood. A cut-off score of 5 is used, insofar that participants with a score more than five likely have depression.

SECONDARY OUTCOMES:
Longterm visuo-spatial memory performance assessed with Starry Night | 1-month follow-up
  Participants are asked to complete the 20-min gamified visuo-spatial memory task, Starry Night, in which they need to remember the shape and location of different, complex patterns.
Quality of life assessed with the QoL Ladder | 1-month follow-up
  Participants are asked to rate their quality of life on a scale from 1 to 8, where 1 is the worst and 8 is the best possible quality of life they could realistically have.
Depressive symptoms assessed with the GDS-15 | 1-month follow-up
  Participants are asked to fill out the GDS-15.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob U Blicher, Professor, Principal Investigator — Aalborg University Hospital
Locations (1):
- Dept. of Neurology, Aalborg University Hospital, Aalborg, North Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT06399978/ICF_000.pdf